CLINICAL TRIAL: NCT03619317
Title: Identification of Chemo and Radiation Induced Systolic and Diastolic Myocardial Dysfunction in Patients With Cancer in Oesophagus and Gastroesophagael Junction - a Prospective Study
Brief Title: Impact of Cancer Therapy on Myocardial Function in Patients With Esophagus Cancer
Acronym: Heartcheck
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Steen Hvitfeldt Poulsen, Associate Professor, MD, Ph.D., DMSci, Aarhus University Hospital Skejby
Other Study IDs: 1-16-02-189-18
Record Dates: First submitted 2018-06-03; First posted 2018-08-07 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cancer of Esophagus
Keywords: Heartdisease; Radiation; Chemoradiotherapy; cardiovascular disease
MeSH Terms: conditions — Esophageal Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer esophagus and gastroesophageal junction: EGEJ cancer patients referred to combined therapy of chemoRT and surgery can be included.

SUMMARY:
Introduction: Patients with cancer in esophagus and gastroesophageal junction (EGEJ) treated with chemoradiotherapy (chemoRT) have increased risk of cardiovascular disease. EGEJ patients often have frailty and pre-existing cardiovascular disease. This may disqualify them for standard trimodal curative treatment and offer surgery alone, chemoRT alone or palliative treatment only. The current understanding of radiation induced heart disease (RIHD) in EGEJ patients is limited. Hence, there is a need for additional studies. Especially on myocardial function during and after chemoRT as congestive heart failure is a serious complication associated with increased morbidity and mortality. Proton-based radiation therapy (RT) is a new alternative to standard photon-based radiation therapy, that is likely to reduce the risk of cardiovascular complications.

Hypothesis: Treatment with chemoRT might induce myocardial dysfunction, symptoms of heart failure and decreased physical performance in patients with EGEJ Cancer.

The aim: Is to investigate the influence on chemoRT on myocardial function in EGEJ patients and evaluate the cardiac prognosis and eventually identify potential high-risk patients who might benefit from proton-based RT instead of the current photon-based RT.

Method: From power calculation the investigators plan to include 56 patients with EGEJ cancer during a period of two years. Inclusions criteria: biopsy verified EGEJ cancer supported by findings from gastroscopy, PET CT scan and with the final diagnosis locally advanced, non-metastatic. The patients will be examined with serial cardiac investigations to evaluate if they develop impairment of the heart function during or after chemoRT. The investigations include; electrocardiogram, cardiac biomarkers, echocardiography and cardio pulmonary exercise test. The examinations will be performed at study entry (baseline) and after six weeks and again after six months.

DETAILED DESCRIPTION:
Background:

Patients with cancer in the esophagus and gastroesophageal junction (EGEJ) treated with chemoradiotherapy (chemoRT) have increased risk of cardiovascular disease. Both chemotherapy and radiotherapy have been reported to be associated with increased cardiovascular morbidity. Still, there is a survival benefit due to multimodal treatment and a careful patient selection. Radiation induced heart disease (RIHD) may include pericarditis, systolic and diastolic myocardial dysfunction, coronary heart disease, valvular heart disease and conduction abnormalities. Standard treatment of locally advanced EGEJ cancer today consists of neoadjuvant chemoRT followed by surgery or chemoRT alone. Elderly patients with frailty and pre-existing cardiovascular disease are in general not offered surgery but might be candidates for treatment with chemoRT alone, still with curative intent. However, the current understanding of RIHD in EGEJ patients is limited as data are sparse. In Sweden a single study has shown that chemoRT might potentially induce acute impairment of both systolic and especially diastolic left ventricular function. The lack of more substantial evidence leaves room for variation in clinical practice. Hence, there is a need for additional studies to provide more insights into the risk of RIHD, in particular on myocardial function during and after chemoRT as congestive heart failure is a serious complication associated with increased morbidity and mortality. Proton-based radiation therapy (RT) is a new alternative to standard photon-based radiation therapy, which reduces the radiation dose to the heart and subsequent risks of cardiovascular complications. However, the availability of proton therapy is still relatively limited for the general EGEJ population, and the indication for proton based RT is not yet evidence based. It is crucial to evaluate risk of heart failure during and after standard chemoRT and to identify potential high-risk patients who might benefit from proton therapy instead of the current standard therapy.

Hypothesis:

Treatment with chemoRT might induce myocardial dysfunction, symptoms of heart failure and decreased physical performance in patients with EGEJ Cancer.

The aim is:

* to identify systolic and diastolic myocardial dysfunction at rest and during peak exercise with advanced non-invasive imaging (echocardiography) following chemoRT.
* to evaluate if baseline myocardial biomarkers (Troponin T (TNT) and N-terminal pro b-type natriuretic peptide (NT-pro-BNP)) and risk factors (diabetes, smoking, hypertension, dyslipidemia) can predict development of myocardial dysfunction.
* to detect whether exercise echocardiography compared to resting echocardiography can identify additional patients with myocardial dysfunction following chemoRT.
* to examine whether development of myocardial dysfunction in EGEJ patients will be reflected in impairment of psychical capacity evaluated by cardiac pulmonary exercise test with assessment of maximal oxygen consumption.
* to evaluate if baseline symptoms classification with clinical frailty score and New York Heart Association (NYHA) and can predict development of myocardial dysfunction.

Method:

Design:

A prospective observational study of patients with EGEJ cancer. Fifty-six patients will be enrolled during a period of 18 months. For the individual patient the heart check investigations will be performed within six months and follow up in general is until 5 years.

After informed consent in the Department of Oncology, the patients will be examined with heart investigations (ECG, Echocardiography rest/exercise and CPX test) in the Department of Cardiology before they start oncologic treatment (baseline) after 6 weeks and again after 6 months.

Clinical frailty, risk factors and cardiac symptoms will be evaluated from structured interview at follow-ups. The investigators will use validated models for graduating risk factors, clinical frailty and shortness of breath (NYHA classification). The patients will serve as own controls comparing the baseline findings with the findings thereafter.

The heart investigations:

Electrocardiogram (ECG): Is made to detect ST-segment depression, elevation or negative T-waves, LV strain or arrhythmias.

Blood samples (Cardiac biomarkers): TNT to detect myocyte necrosis and NT-pro-BNP to detect myocardial dysfunction and lipids to be used in risk evaluation.

3D echocardiography at rest and during exercise: Two-and three-dimensional Doppler echocardiography is used to evaluate Left ventricular (LV) systolic and diastolic function.

LV systolic function is evaluated by 3D echocardiography estimated ejection fraction (LVEF) and by 2D global longitudinal strain (GLS), which is a sensitive marker of myocardial function beyond LVEF. The test will be performed at rest and at peak exercise using a semi-supine ergometer bicycle. Determination of LV contractile reserve capacity is evaluated by the difference in GLS and LVEF at rest and at peak exercise. Myocardial systolic reserve capacity in other cardiac diseases has demonstrated to be a significant marker of functional capacity.

LV diastolic function is evaluated by left atrial volume and pulsed and tissue-Doppler parameters according to current guidelines by the European Society of Cardiology.

Cardio pulmonary exercise (CPX) test:

Maximum oxygen uptake (VO2 max) from a cardio pulmonary test is gold standard to measure the physically capacity of patients and is known to add prognostic information in patients with heart failure independently of etiology. The patient will be placed on a semi-supine special designed bicycle with simultaneous determination of VO2 during increasing watts. Hemodynamic parameters as pulse, blood pressure and ECG will be measured continuously. Echocardiography will be performed at rest and during peak exercise

ELIGIBILITY:
Inclusion Criteria:

* Biopsy verified EGEJ cancer verified by gastroscopy, biopsy and PET/CT scan.
* The final diagnosis must be locally advanced, non-metastatic as determined at a multidisciplinary team conference.
* Patients referred to curative treatment with preoperative or definitive chemo- and radiotherapy.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age < 18 years
  * Patients not being able to give informed consent (decided by the investigator).
  * Patients not being able to understand Danish language.
  * Acute myocardial infarct within the last 6 months.
  * Present clinical severe heart valve disease and/or congestive heart failure with left ejection fraction < 25 %.
  * Patients with prior thoracic radiation and overlapping RT fields.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
• Left ventricular systolic function estimated by 2D longitudinal strain (GLS) and ejection fraction (EF) at rest and peak exercise | From Baseline till 6 weeks after.
  where a decrease of peak GLS of 10 % is considered clinical significant.

SECONDARY OUTCOMES:
• Change of NT-pro-BNP | From Baseline till 6 weeks after.
  with a double increase provided that serum level is above >300 pmol/L after ChemoRT provided e-GFR >30 ml/min.
• Change in TNT | From Baseline till 6 weeks after.
  2 x upper normal value = >28 ng/l provided that Estimated glomerular filtration rate >50 ml/min.
• Change of peak VO2 | From Baseline till 6 weeks after.
  of 10% ml/kg/min after chemoRT compared to baseline.
• Change in diastolic function | From Baseline till 6 weeks after.
  defined as an increase of at least one diastolic grade
• Admission to hospital with clinical heart failure. | Baseline, after 4 weeks and 6 months.
  To investigate if the have had heart related admission to hospital
• Dead - not cancer related. | From Baseline till 6 weeks after.
  Dead that is not related to the cancer diagnosis
• Increased use of diuretics compared to baseline | Baseline, after 4 weeks and 6 months.
  accumulated use of thiazide, loop or aldosterone antagonists
• Change in use of ace-inhibitors, betablockers, digoxin and hydralazine compared to baseline. | From Baseline till 6 weeks after.
  Increased use of the drugs mentioned
Left ventricular systolic function estimated by 2D longitudinal strain (GLS) and ejection fraction (EF) at rest and peak exercise | From Baseline till 6 weeks after.
  where a decrease of EF 5 % (absolute) is considered clinical significant.

CONTACTS AND LOCATIONS:
Overall Officials: Steen H Poulsen, MD phd DMSci, Principal Investigator — Aarhus University Hopital, Skejby, Department of Cardiology
Locations (1):
- University Hospital of Aarhus, Department of Cardiology, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nielsen KM, Offersen BV, Nielsen HM, Vaage-Nilsen M, Yusuf SW. Short and long term radiation induced cardiovascular disease in patients with cancer. Clin Cardiol. 2017 Apr;40(4):255-261. doi: 10.1002/clc.22634. Epub 2017 Jan 31. PMID 28139844
- [Background] Madan R, Matalon S, Vivero M. Spectrum of Smoking-related Lung Diseases: Imaging Review and Update. J Thorac Imaging. 2016 Mar;31(2):78-91. doi: 10.1097/RTI.0000000000000185. PMID 26479130
- [Background] Beukema JC, van Luijk P, Widder J, Langendijk JA, Muijs CT. Is cardiac toxicity a relevant issue in the radiation treatment of esophageal cancer? Radiother Oncol. 2015 Jan;114(1):85-90. doi: 10.1016/j.radonc.2014.11.037. Epub 2014 Dec 30. PMID 25554226
- [Background] Lund M, Alexandersson von Dobeln G, Nilsson M, Winter R, Lundell L, Tsai JA, Kalman S. Effects on heart function of neoadjuvant chemotherapy and chemoradiotherapy in patients with cancer in the esophagus or gastroesophageal junction - a prospective cohort pilot study within a randomized clinical trial. Radiat Oncol. 2015 Jan 13;10:16. doi: 10.1186/s13014-014-0310-7. PMID 25582305
- [Background] Clemmensen TS, Eiskjaer H, Molgaard H, Larsen AH, Soerensen J, Andersen NF, Tolbod LP, Harms HJ, Poulsen SH. Abnormal Coronary Flow Velocity Reserve and Decreased Myocardial Contractile Reserve Are Main Factors in Relation to Physical Exercise Capacity in Cardiac Amyloidosis. J Am Soc Echocardiogr. 2018 Jan;31(1):71-78. doi: 10.1016/j.echo.2017.09.007. Epub 2017 Oct 27. PMID 29111120
- [Background] Chuong MD, Hallemeier CL, Jabbour SK, Yu J, Badiyan S, Merrell KW, Mishra MV, Li H, Verma V, Lin SH. Improving Outcomes for Esophageal Cancer using Proton Beam Therapy. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):488-497. doi: 10.1016/j.ijrobp.2015.11.043. Epub 2015 Dec 14. PMID 27084662
- [Background] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Background] Xi M, Xu C, Liao Z, Chang JY, Gomez DR, Jeter M, Cox JD, Komaki R, Mehran R, Blum MA, Hofstetter WL, Maru DM, Bhutani MS, Lee JH, Weston B, Ajani JA, Lin SH. Comparative Outcomes After Definitive Chemoradiotherapy Using Proton Beam Therapy Versus Intensity Modulated Radiation Therapy for Esophageal Cancer: A Retrospective, Single-Institutional Analysis. Int J Radiat Oncol Biol Phys. 2017 Nov 1;99(3):667-676. doi: 10.1016/j.ijrobp.2017.06.2450. Epub 2017 Jun 27. PMID 29280461
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Alexandru Popescu B, Waggoner AD; Houston, Texas; Oslo, Norway; Phoenix, Arizona; Nashville, Tennessee; Hamilton, Ontario, Canada; Uppsala, Sweden; Ghent and Liege, Belgium; Cleveland, Ohio; Novara, Italy; Rochester, Minnesota; Bucharest, Romania; and St. Louis, Missouri. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1321-1360. doi: 10.1093/ehjci/jew082. Epub 2016 Jul 15. No abstract available. PMID 27422899
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Derived] Astrup Sondergaard MM, Nordsmark M, Sloth Moller D, Melgaard Nielsen K, Poulsen SH. Reduction in myocardial function and oxygen consumption after chemoradiotherapy in patients with esophageal cancer. Acta Oncol. 2022 May;61(5):566-574. doi: 10.1080/0284186X.2022.2048068. Epub 2022 Mar 15. PMID 35289694
- [Derived] Sondergaard MMA, Nordsmark M, Nielsen KM, Poulsen SH. Cardiovascular Burden and Adverse Events in Patients With Esophageal Cancer Treated With Chemoradiation for Curative Intent. JACC CardioOncol. 2021 Dec 21;3(5):711-721. doi: 10.1016/j.jaccao.2021.10.002. eCollection 2021 Dec. PMID 34988480